CLINICAL TRIAL: NCT04625062
Title: Comparing Traditional and Biofeedback Treatment for Residual Speech Errors Via Telepractice
Brief Title: Comparing Traditional and Biofeedback Telepractice Treatment for Residual Speech Errors
Acronym: C-RESULTS TPT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Syracuse University (Other); Montclair State University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C-RESULTS-TPT; R01DC017476 (NIH)
Record Dates: First submitted 2020-09-08; First posted 2020-11-12 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2020-11

CONDITIONS: Speech Sound Disorder
Keywords: speech; articulation; motor development
MeSH Terms: conditions — Speech Sound Disorder; Speech

STUDY DESIGN:
Intervention Model Description: In this within-subjects single-case randomization design, each participant will receive an equal number of sessions of visual-acoustic biofeedback and traditional treatment (n = 10 each), with randomized allocation of treatment types to individual sessions. Randomization will be blocked, with each week of treatment serving as a block; within each week/block, one session will be randomly assigned to feature visual-acoustic and one to feature traditional treatment.
Who Masked: Outcomes Assessor
Masking Description: All perceptual ratings will be obtained from blinded, naive listeners recruited through online crowdsourcing. Following protocols refined in previous published research, binary rating responses will be aggregated over at least 9 unique listeners per token.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual-acoustic biofeedback (Experimental): Visual- acoustic biofeedback treatment (behavioral) administered via telepractice
  Interventions: Behavioral: Visual-acoustic biofeedback
- Motor-based treatment (Experimental): Motor-based articulation treatment administered via telepractice
  Interventions: Behavioral: Motor-based treatment

INTERVENTIONS:
Behavioral: Visual-acoustic biofeedback — In visual-acoustic biofeedback treatment, participants view a dynamic display of the speech signal in the form of a real-time LPC (Linear Predictive Coding) spectrum. Because correct vs incorrect productions of /r/ contrast acoustically in the frequency of the third formant (F3), participants were cued to make their real-time LPC spectrum match a visual target characterized by a low F3 frequency.
  Arms: Visual-acoustic biofeedback
Behavioral: Motor-based treatment — Motor-based articulation treatment involves providing auditory models and verbal descriptions of correct articulator placement, then cueing repetitive motor practice. Images and diagrams of the vocal tract were used as visual aids; however, no real-time visual display of articulatory or acoustic information will be made available.
  Arms: Motor-based treatment

SUMMARY:
This study aims to evaluate the relative efficacy of biofeedback and traditional treatment for residual speech errors when both are delivered via telepractice. In a single-case randomization design, up to eight children with RSE will receive both visual-acoustic biofeedback and traditional treatment via telepractice. Acoustic measures of within-session change will be compared across sessions randomly assigned to each condition. It is hypothesized that participants will exhibit a clinically significant overall treatment response and that short-term measures of change will indicate that biofeedback is associated with larger increments of progress than traditional treatment.

DETAILED DESCRIPTION:
The COVID-19 crisis has forced speech-language pathologists to migrate from in-person delivery of speech treatment services to remote delivery via telepractice. This study will compare the efficacy of visual-acoustic biofeedback treatment versus non-biofeedback treatment in this setting. Specifically, participants will receive both visual-acoustic biofeedback treatment and non-biofeedback treatment via telepractice (Zoom call with screen-sharing) in a single-case randomization design. The hypothesis of interest is that sessions featuring visual-acoustic biofeedback will be associated with larger short-term gains than sessions featuring non-biofeedback treatment. To test this hypothesis, the study team will recruit up to 8 participants who will receive an initial treatment orientation followed by an equal dose of both types of treatment (10 sessions of visual-acoustic biofeedback and 10 sessions of non-biofeedback treatment). Participants will complete approximately two sessions per week via telepractice; each week will feature one session of each type, randomly ordered. They will also complete 4 pre-treatment baseline sessions and 3 post-treatment maintenance sessions to evaluate the overall magnitude of change over the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 9;0 and 15;11 years of age at the time of enrollment.
* Must speak English as the dominant language (i.e., must have begun learning English by age 2, per parent report).
* Must speak a rhotic dialect of English.
* Must pass a brief examination of oral structure and function.
* Must exhibit less than thirty percent accuracy, based on trained listener ratings, on a probe list eliciting /r/ in various phonetic contexts at the word level.

Exclusion Criteria:

* Must not receive a T score more than 1.3 standard deviations (SD) below the mean on the Wechsler Abbreviated Scale of Intelligence-2 (WASI-2) Matrix Reasoning.
* Must not receive a scaled score below 6 on the CELF-5 Recalling Sentences or Formulated Sentences subtests.
* Must not have history of sensorineural hearing loss or failed infant hearing screening.
* Must not have an existing diagnosis of developmental disability, major neurobehavioral syndrome such as cerebral palsy, Down Syndrome, or Autism Spectrum Disorder, or major neural disorder (e.g., epilepsy, agenesis of the corpus callosum) or insult (e.g., traumatic brain injury, stroke, or tumor resection).
* Must not show clinically significant signs of apraxia of speech or dysarthria.
* Must not have major orthodontia that could interfere with tongue-palate contact.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Montclair State University, Bloomfield, New Jersey
  - Syracuse University, Syracuse, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dugan SH, Silbert N, McAllister T, Preston JL, Sotto C, Boyce SE. Modelling category goodness judgments in children with residual sound errors. Clin Linguist Phon. 2019;33(4):295-315. doi: 10.1080/02699206.2018.1477834. Epub 2018 May 24. PMID 29792525
- [Background] Campbell H, Harel D, Hitchcock E, McAllister Byun T. Selecting an acoustic correlate for automated measurement of American English rhotic production in children. Int J Speech Lang Pathol. 2018 Nov;20(6):635-643. doi: 10.1080/17549507.2017.1359334. Epub 2017 Aug 10. PMID 28795872
- [Background] Campbell H, McAllister Byun T. Deriving individualised /r/ targets from the acoustics of children's non-rhotic vowels. Clin Linguist Phon. 2018;32(1):70-87. doi: 10.1080/02699206.2017.1330898. Epub 2017 Jul 13. PMID 28703653
- [Background] McAllister Byun T. Efficacy of Visual-Acoustic Biofeedback Intervention for Residual Rhotic Errors: A Single-Subject Randomization Study. J Speech Lang Hear Res. 2017 May 24;60(5):1175-1193. doi: 10.1044/2016_JSLHR-S-16-0038. PMID 28389677
- [Background] McAllister Byun T, Tiede M. Perception-production relations in later development of American English rhotics. PLoS One. 2017 Feb 16;12(2):e0172022. doi: 10.1371/journal.pone.0172022. eCollection 2017. PMID 28207800
- [Background] McAllister Byun T, Campbell H. Differential Effects of Visual-Acoustic Biofeedback Intervention for Residual Speech Errors. Front Hum Neurosci. 2016 Nov 11;10:567. doi: 10.3389/fnhum.2016.00567. eCollection 2016. PMID 27891084
- [Background] McAllister Byun T, Halpin PF, Szeredi D. Online crowdsourcing for efficient rating of speech: a validation study. J Commun Disord. 2015 Jan-Feb;53:70-83. doi: 10.1016/j.jcomdis.2014.11.003. Epub 2014 Dec 15. PMID 25578293
- [Background] Harel D, Hitchcock ER, Szeredi D, Ortiz J, McAllister Byun T. Finding the experts in the crowd: Validity and reliability of crowdsourced measures of children's gradient speech contrasts. Clin Linguist Phon. 2017;31(1):104-117. doi: 10.3109/02699206.2016.1174306. Epub 2016 Jun 7. PMID 27267258
- [Background] Hitchcock ER, Harel D, Byun TM. Social, Emotional, and Academic Impact of Residual Speech Errors in School-Aged Children: A Survey Study. Semin Speech Lang. 2015 Nov;36(4):283-94. doi: 10.1055/s-0035-1562911. Epub 2015 Oct 12. PMID 26458203
- [Background] Byun TM, Hitchcock ER. Investigating the use of traditional and spectral biofeedback approaches to intervention for /r/ misarticulation. Am J Speech Lang Pathol. 2012 Aug;21(3):207-21. doi: 10.1044/1058-0360(2012/11-0083). Epub 2012 Mar 21. PMID 22442281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Institutional review board approval was obtained from the Biomedical Research Alliance of New York (BRANY, protocol number 18-10-393). Participants, who could come from anywhere in the US, were recruited through recruitment flyers, listserv announcements, and social media posts.
Pre-assignment Details: This study used a within-subjects design. Each participant received both treatment conditions, with sessions randomly assigned to feature one condition or the other (n = 10 sessions in each condition).
Units Other Than Participants: Sessions
Groups:
- Visual-acoustic Biofeedback: Visual-acoustic biofeedback: In visual-acoustic biofeedback treatment, the elements of motor-based treatment (i.e., auditory models and verbal descriptions of articulator placement) are enhanced with a dynamic display of the speech signal in the form of the real-time LPC (Linear Predictive Coding) spectrum. Because correct vs incorrect productions of /r/ contrast acoustically in the frequency of the third formant (F3), participants will be cued to make their real-time LPC spectrum match a visual target characterized by a low F3 frequency. They will be encouraged to attend to the visual display while adjusting the placement of their articulators and observing how those adjustments impact F3. All treatment will be provided over video calls. All participants completed 10 sessions in the visual-acoustic biofeedback condition.
- Motor-based Treatment: Motor-based treatment: Motor-based articulation treatment involves providing auditory models and verbal descriptions of correct articulator placement, then cueing repetitive motor practice. Images and diagrams of the vocal tract will be used as visual aids; however, no real-time visual display of articulatory or acoustic information will be made available. All treatment will be provided over video calls. All participants completed 10 sessions in the motor-based treatment condition.
Period: Overall Study
Arm/Group | Visual-acoustic Biofeedback | Motor-based Treatment
Started | 7; 10 Sessions | 7; 10 Sessions
Completed | 7; 10 Sessions | 7; 10 Sessions
Not Completed | 0; 0 Sessions | 0; 0 Sessions

BASELINE CHARACTERISTICS:
Population: Note that, due to the within-subject design of the study, participants in Condition 1 are the same as participants in Condition 2.
Groups:
- Visual-acoustic Biofeedback and Motor-based Treatment: This study used a within-subjects randomization design. Each participant received both treatment conditions, with sessions randomly assigned to feature one condition or the other.
  Visual-acoustic biofeedback treatment (behavioral) administered via telepractice
  Visual-acoustic biofeedback: In visual-acoustic biofeedback treatment, the elements of motor-based treatment (i.e., auditory models and verbal descriptions of articulator placement) are enhanced with a dynamic display of the speech signal in the form of the real-time LPC (Linear Predictive Coding) spectrum. Because correct vs incorrect productions of /r/ contrast acoustically in the frequency of the third formant (F3), participants will be cued to make their real-time LPC spectrum match a visual target characterized by a low F3 frequency. They will be encouraged to attend to the visual display while adjusting the placement of their articulators and observing how those adjustments impact F3. All treatment will be provided over video calls.
  Motor-based articulation treatment administered via telepractice
  Motor-based treatment: Motor-based articulation treatment involves providing auditory models and verbal descriptions of correct articulator placement, then cueing repetitive motor practice. Images and diagrams of the vocal tract will be used as visual aids; however, no real-time visual display of articulatory or acoustic information will be made available. All treatment will be provided over video calls.
Arm/Group | Visual-acoustic Biofeedback and Motor-based Treatment
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: months] | 132 (21.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
Percent /r/ sounds correct [Mean (Standard Deviation); unit: Percentage words rated correct] | 19.4 (18.6)

OUTCOME MEASURES:

1. Primary Outcome: Within-session Change in Percentage of "Correct" Ratings by Blinded Naive Listeners for /r/ Sounds Produced in Word Probes
Description: To assess /r/ production accuracy, participants read probe lists eliciting 25 utterances of /r/ in various phonetic contexts at the start and end of each treatment session. Recorded probe words are presented in randomized order for binary rating (correct/incorrect) by naive listeners who are blind to treatment condition and time point; the accuracy of each token is quantified as the percentage of "correct" ratings across 9 blinded listeners. We then compute the mean percent correct ratings for each probe; the change in this value from pre to post session ("within-session change") is our outcome measure of interest. Summary statistics report the mean and standard deviation of within-session change for each treatment condition, pooled across participants and sessions. This Outcome Measure is assessed using a two-tailed paired-samples t-test comparing mean change in percent correct for each treatment condition across subjects. Outcomes are evaluated relative to a superiority criterion.
Time Frame: Change in word probe accuracy was measured in each treatment session, which were administered over ten weeks.
Population: Note that this study used a within-subjects design. Each participant received both treatment conditions, with individual sessions randomly assigned to feature one condition or the other.
Measure: Mean (Standard Deviation); unit: Percent correct
Units Other Than Participants: Sessions
Groups:
- Condition 1: Visual-acoustic Biofeedback: Visual-acoustic biofeedback treatment (behavioral) administered via telepractice
  Visual-acoustic biofeedback: In visual-acoustic biofeedback treatment, the elements of motor- based treatment (i.e., auditory models and verbal descriptions of articulator placement) are enhanced with a dynamic display of the speech signal in the form of the real-time LPC (Linear Predictive Coding) spectrum. Because correct vs incorrect productions of /r/ contrast acoustically in the frequency of the third formant (F3), participants will be cued to make their real-time LPC spectrum match a visual target characterized by a low F3 frequency. They will be encouraged to attend to the visual display while adjusting the placement of their articulators and observing how those adjustments impact F3. All treatment will be provided over video calls.
- Condition 2: Motor-based Treatment: Motor-based articulation treatment administered via telepractice
  Motor-based treatment: Motor-based articulation treatment involves providing auditory models and verbal descriptions of correct articulator placement, then cueing repetitive motor practice. Images and diagrams of the vocal tract will be used as visual aids; however, no real-time visual display of articulatory or acoustic information will be made available. All treatment will be provided over video calls.
Arm/Group | Condition 1: Visual-acoustic Biofeedback | Condition 2: Motor-based Treatment
Number analyzed (Participants) | 7 | 7
Number analyzed (Sessions) | 10 | 10
Percent correct | 1.4 (8.3) | 1.9 (9.6)
Statistical Analysis 1: Comparison: Condition 1: Visual-acoustic Biofeedback vs Condition 2: Motor-based Treatment; Test type: Superiority; p = .72, paired t-test, two-tailed; df = 6; Mean Difference (Final Values) = .49 — Traditional treatment condition - biofeedback treatment condition

ADVERSE EVENTS:
Time Frame: 6.5 months
Description: The definition of adverse event and serious adverse event used to collect adverse event information does not differ from that of clinicaltrials.gov.
Groups:
- Condition 1: Visual-acoustic Biofeedback: Visual-acoustic biofeedback treatment (behavioral) administered via telepractice
  Visual-acoustic biofeedback: In visual-acoustic biofeedback treatment, the elements of motor-based treatment (i.e., auditory models and verbal descriptions of articulator placement) are enhanced with a dynamic display of the speech signal in the form of the real-time LPC spectrum. All treatment will be provided over video calls.
Arm/Group | Condition 1: Visual-acoustic Biofeedback | Condition 2: Motor-based Treatment
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
Single-case randomization designs are limited in that gains from one treatment condition may carry over to the next.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT04625062/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT04625062/SAP_001.pdf